CLINICAL TRIAL: NCT01207843
Title: Verbesserung Der Radiologischen Diagnose Von Hepatolienaler Candidiasis während Der Therapie Der Leukämie
Brief Title: Optimized Radiological Diagnosis of Hepatic Candidiasis During the Treatment of Acute Leukemias
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: idr-3d-001
Record Dates: First submitted 2010-09-21; First posted 2010-09-23 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Leukemia; Infection
Keywords: Computed tomography
MeSH Terms: conditions — Leukemia; Infections | interventions — X-Rays

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Imaging — CT image validation and lesion measurement, as well as comparison of different CT phases

SUMMARY:
Hepatic candidiasis is a frequent complication in patients receiving intensive chemotherapy for acute leukemia. Hepatic lesions may be detected by computerized tomographic (CT) scans, but there is no standardized CT protocol for the diagnosis and follow-up of hepatic candidiasis.

The investigators compared the size of the fungal lesions in the chest and abdomen CT. The current analysis aimed to increase the value of CT for the diagnosis and the follow-up of hepatic candidiasis in daily routine.

ELIGIBILITY:
Inclusion criteria:

* Chest and Abdomen CT with fungal lesion in patients with leukemia

Exclusion criteria:

* Other liver pathologies

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with suspected hepatolienal candidiasis.
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2009-10; Primary Completion 2011-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The primary end-point was IFI according to the EORTC/MSG 2008 definitions and bacteraemia | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Frauenfelder, MD, Principal Investigator — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland